CLINICAL TRIAL: NCT07130448
Title: The Relation of Albumin/Globulin Ratio and Platelet/Albumin Ratio to Lupus Nephritis in Upper Egypt ( Single Center Study)
Brief Title: The Relation of Albumin/Globulin Ratio and Platelet/Albumin Ratio to Lupus Nephritis
Status: Not yet recruiting | Type: Observational
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Mina Maged William, Doctor, Assiut University
Other Study IDs: Lupus Nephritis biomarkers
Record Dates: First submitted 2025-08-10; First posted 2025-08-19 (Actual); Last update posted 2025-08-19 (Actual); Status verified 2025-08

CONDITIONS: Lupus Nephritis (LN); SLE - Systemic Lupus Erythematosus; Biomarkers
MeSH Terms: conditions — Lupus Nephritis; Lupus Erythematosus, Systemic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Albumin/globulin ratio and platelet/albumin ratio as a predictive non-invasive biomarker for lupus nephritis (LN) presence and severity

DETAILED DESCRIPTION:
Lupus nephritis (LN) is one of the most frequent and severe manifestations of systemic lupus erythematosus (SLE) and serves as a major predictor of poor prognosis . Delayed diagnosis significantly increases the risk of renal insufficiency and progression to end-stage renal disease (ESRD) . Conventional laboratory markers-such as proteinuria, urine protein-to-creatinine ratio, creatinine clearance, anti-double-stranded DNA (anti-dsDNA) antibodies, and complement levels-are commonly used to assess LN . However, these markers often lack sufficient sensitivity and specificity for early diagnosis and disease monitoring .This limitation has prompted interest in identifying reliable, non-invasive, and cost-effective biomarkers for LN. The albumin/globulin (A/G) ratio is one such biomarker, reflecting systemic inflammation and immune dysregulation. In SLE, inflammation or proteinuria often leads to hypoalbuminemia, while increased immunoglobulin production elevates globulin levels, reducing the A/G ratio. Lower ratios have been associated with increased disease activity and organ damage .

Another emerging marker is the platelet/albumin (P/A) ratio, which integrates inflammatory status with nutritional and renal function indicators. It has demonstrated prognostic value in diabetes mellitus ,cardiovascular, hepatic, and autoimmune conditions .Despite their promise, these biomarkers have not been adequately studied in Egyptian LN patients. Given that regional and demographic variations may influence disease expression, evaluating these ratios in Upper Egypt may provide clinically relevant insights and inform local disease management strategies.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 18 years or older diagnosed as SLE according to 2019 ACR/EULAR classification criteria and with lupus nephritis (LN) according to the ACR criteria.
* Patients with available baseline laboratory investigations and renal biopsy.

Exclusion Criteria:

* Patients with chronic liver disease, hematological disorders, or malignancies affecting albumin/globulin ratio or platelet counts.
* Patients on nephrotoxic medications not related to SLE management.
* Recent infections or acute inflammatory conditions.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Aged ≥18 years.
  * SLE patients fulfilling the SLE International Collaborating Clinics (SLICC) - ----classification criteria and matched controls.
  * Patients cooperative and can answer questions.
  * Patients who are able and willing to give written informed consent.
Sampling Method: Non-Probability Sample
Enrollment: 120 (Estimated)
Dates: Start 2025-09 (Estimated); Primary Completion 2026-09 (Estimated); Study Completion 2026-10 (Estimated)

PRIMARY OUTCOMES:
Association of Albumin/Globulin (A/G) and Platelet/ Albumin (P/A) ratios with the presence of lupus nephritis | baseline
  unit of measurments : ratios (no units )
Compare the Albumin/Globulin (A/G) and Platelet/Albumin (P/A) ratios between different classes of lupus nephritis | baseline
  unite of measurments : ratios (no units )

SECONDARY OUTCOMES:
• Correlation of A/G and P/A ratios with lupus nephritis class, 24-hour urine protein or urine protein/creatinine ratio, Serum creatinine and eGFR. | baseline
• Predictive value of A/G and P/A ratios for renal involvement: Using logistic regression or ROC curve analysis to assess whether these ratios can predict the presence of nephritis. | baseline

REFERENCES:
- [Background] Leng L, Shen J, Li L, Li J, Li X, Liu D. Nonlinear association between platelet to albumin ratio and disease activity in patients with early rheumatoid arthritis. Sci Rep. 2024 Nov 7;14(1):27112. doi: 10.1038/s41598-024-78582-1. PMID 39511276
- [Background] Cao SL, Zhang GQ, Li J, Bao L, Lan XM, Jin QP, Luo HY, E J, Li B, Ma D, Bao X, Zheng YL. Platelet-to-albumin ratio is a potential biomarker for predicting diabetic nephropathy in patients with type 2 diabetes. Biomark Med. 2023 Oct;17(20):841-848. doi: 10.2217/bmm-2023-0527. Epub 2024 Jan 5. PMID 38180339
- [Background] Hao P, Feng S, Suo M, Wang S, Wu X. Platelet to albumin ratio: A risk factor related to prognosis in patients with non-ST-segment elevation acute coronary syndrome undergoing percutaneous coronary intervention. Int J Cardiol. 2024 Jan 15;395:131588. doi: 10.1016/j.ijcard.2023.131588. Epub 2023 Nov 19. PMID 37989451
- [Background] Liu M, Li X, Huang Y, Huang Z, Huang Q. Albumin to globulin ratio (AGR) in systemic lupus erythematosus: correlation with disease activity. J Int Med Res. 2024 Apr;52(4):3000605241244761. doi: 10.1177/03000605241244761. PMID 38661083
- [Background] Mok CC. Biomarkers for lupus nephritis: a critical appraisal. J Biomed Biotechnol. 2010;2010:638413. doi: 10.1155/2010/638413. Epub 2010 Apr 19. PMID 20414362
- [Background] Faurschou M, Starklint H, Halberg P, Jacobsen S. Prognostic factors in lupus nephritis: diagnostic and therapeutic delay increases the risk of terminal renal failure. J Rheumatol. 2006 Aug;33(8):1563-9. PMID 16881113
- [Background] Dumestre-Perard C, Clavarino G, Colliard S, Cesbron JY, Thielens NM. Antibodies targeting circulating protective molecules in lupus nephritis: Interest as serological biomarkers. Autoimmun Rev. 2018 Sep;17(9):890-899. doi: 10.1016/j.autrev.2018.03.013. Epub 2018 Jul 29. PMID 30009962